CLINICAL TRIAL: NCT02207049
Title: The Effect of Snack Consumption on Energy Intake in Preschoolers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9564 B
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Energy Intake; Snacks; Children, Preschool
MeSH Terms: interventions — Snacks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Three Meals (TM) (Active Comparator): Preschoolers will be provided their caloric needs within three meals.
  Interventions: Behavioral: No Snacking
- Meal plus Snack (M+S) (Active Comparator): Preschoolers will be provided three meals and two snacks, with total amount of food provided in the day the same as the Three Meal (TM) arm.
  Interventions: Behavioral: Snacking
- Three Meal plus Snack (TM+S) (Active Comparator): Preschoolers will be provided three meals and two snacks with total amount provided in the meals equal to the Three Meal (TM) arm and total amount provided in the snacks equal to Meal plus Snacks (M+S) arm.
  Interventions: Behavioral: Snacking

INTERVENTIONS:
Behavioral: Snacking — Snacks will be provided to preschoolers, either as part of total caloric needs or above total caloric needs
  Arms: Meal plus Snack (M+S); Three Meal plus Snack (TM+S)
Behavioral: No Snacking — Caloric needs will be provided to preschoolers within three meals
  Arms: Three Meals (TM)

SUMMARY:
The purpose of this pilot study will be to examine the influence of providing snacks on consumption of overall energy intake in children aged 2-5 years in the Early Learning Center (ELC) at the University of Tennessee.

DETAILED DESCRIPTION:
Providing snacks to children is widely recommended for appetite regulation and assisting with meeting nutritional guidelines.1 Currently, snacks contribute a larger portion of dietary intake in children than in previous years.2,3 Additionally, observational research has found that self-reported, low-nutrient-dense snack consumption, has increased among preschoolers (ages 2-to-6 years) over the past 20 years, leading to an increase of total daily energy intake.3 However, no experimental studies examining the influence of snack intake on energy consumption in children have been conducted.2 Therefore, at this time it is not clear how snacks impact appetite regulation or energy intake, especially in young children.

Thus, the purpose of this pilot study will be to examine the influence of providing snacks on consumption of overall energy intake in children aged 2-5 years in the Early Learning Center (ELC) at the University of Tennessee. Children will be provided with 3-to-5 ad libitum eating occasions over the course of a day for three sessions. To test the effects of providing snacks to preschoolers on consumption of food throughout the day, the food will be provided in three ways in the three different sessions: 1) children will be provided three meals (TM); 2) children will be provided three meals and two snacks, with total amount of food provided in the day the same as TM (M+S); and 3) children will be provided three meals and two snacks with total amount provided in the meals equal to TM and total amount provided in the snacks equal to M+S (TM+S).

Primary Hypothesis:

1) Energy consumed from food and beverages will be greatest during the TM+S session, followed by M+S, and then TM.

ELIGIBILITY:
Inclusion Criteria:

* 3 -to- 5 years of age
* enrolled at the Early Learning Center for the full day program
* have guardian consent to participate
* like the foods served

Exclusion Criteria:

* have allergies or intolerances to the foods being served
* not able to use a spoon
* did not attend all feeding sessions

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Total calories of the food and beverages consumed. | 3 weeks
  Total calories of food and beverage consumed by participants over the 3-week study (with 1 day of food and beverage per week) period will be determined by subtracting pre- and post-consumption weight of the food and beverage provided and multiplied by the energy density of each respective food and beverage.

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A Raynor, PhD, RD, LDN, Principal Investigator — University of Tennesseem Knoxville
Locations (1):
- Healthy Eating and Activity Laboratory, Knoxville, Tennessee, United States

REFERENCES:
- [Background] Allen RE, Myers AL. Nutrition in toddlers. Am Fam Physician. 2006 Nov 1;74(9):1527-32. PMID 17111891
- [Background] Smith-Petersen MN, Larson CB, Cochran W. Local chemotherapy with primary closure of septic wounds by means of drainage and irrigation cannulae : M. N. Smith-Petersen MD (1886-1953), Carroll B. Larson MD, Williams Cochran MD . The 12th president of the AAOS 1943 (MNS-P). Clin Orthop Relat Res. 2008 Jan;466(1):104-12. doi: 10.1007/s11999-007-0023-4. PMID 18196379
- [Background] Ford CN, Slining MM, Popkin BM. Trends in dietary intake among US 2- to 6-year-old children, 1989-2008. J Acad Nutr Diet. 2013 Jan;113(1):35-42. doi: 10.1016/j.jand.2012.08.022. PMID 23260722